CLINICAL TRIAL: NCT01425775
Title: The Effect of Vitamin D Supplementation on Disease Activity Markers in Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, Professor of Rheumatology, University of Alexandria
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: alexmed116618166
Record Dates: First submitted 2011-08-18; First posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; disease activity markers; vitamin D
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator)
  Interventions: Drug: vitamin D 25(OH)D
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: vitamin D 25(OH)D — 2000IU/day for 12 months
  Arms: Vitamin D
Other: Placebo — 2000IU/day of vitamin D will be compared to similar looking tablets of placebo for 12 months
  Arms: Placebo

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic multi-system inflammatory autoimmune disease. Vitamin D has potent immunomodulatory properties that have promoted its potential use in the treatment of autoimmune conditions, including SLE. We assessed vitamin D status in SLE patients and determined alterations in inflammatory, hemostatic markers as well as disease activity before and after vitamin D supplementation.

248 SLE patients were enrolled in this randomized placebo-controlled study. Patients were randomized 2:1 to receive either oral cholecalciferol 2000 IU/day or placebo for 12 months. Outcome measures included assessment of alterations in levels of IL-1, IL-6, IL-18, TNF-alpha, Anti-dsDNA, ANA, fibrinogen and von Willebrand Factor (vWF) before and after 12 months supplementation. Disease activity was measured by the SLEDAI. Vitamin D levels were measured by Liaison immunoassay; (normal 30-100ng/ml). Serum levels between 10-30 ng/ml were classified as vitamin D insufficiency, and levels < 10 ng/ml as vitamin D deficiency.The mean 25(OH) D level at baseline was 19.8 ng/ml in patients compared to 28.7 ng/ml in controls.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women and males of the same body mass index and ethnicity

Exclusion Criteria:

Patients with:

* other inflammatory disorders,
* hepatic disease
* renal disease
* malignant disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Decrease in SLE disease activity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Abou-Raya, MD, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Egypt

REFERENCES:
- [Derived] Abou-Raya A, Abou-Raya S, Helmii M. The effect of vitamin D supplementation on inflammatory and hemostatic markers and disease activity in patients with systemic lupus erythematosus: a randomized placebo-controlled trial. J Rheumatol. 2013 Mar;40(3):265-72. doi: 10.3899/jrheum.111594. Epub 2012 Dec 1. PMID 23204220 (Retraction: PMID 30504482 J Rheumatol. 2018 Dec;45(12):1713)